CLINICAL TRIAL: NCT00410839
Title: Prevention of Atrial Fibrillation Recurrence By An Alpha-Linolenic Enriched Diet - A Pilot Study
Brief Title: Studies of the Prevention of Atrial Fibrillation by ALA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Hospital, Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 99-04 (CPPRB Bordeaux B)
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2006-12-13 (Estimated); Status verified 2004-08

CONDITIONS: Atrial Fibrillation; Diet Therapy
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Procedure: ALA rich diet

SUMMARY:
An alpha-linolenic acid (ALA) rich diet in the Lyon Heart Study reduced sudden cardiac deaths possibly by reducing cardiac arrhythmias and ventricular fibrillation (Lancet 1994). Since then, there has been a growing interest in ALA as a cardioprotective nutrient. Much of the interest has focused on the potential antiarrhythmic effect of ω-3 fatty acids, especially the longer chain ω-3 fatty acids, DHA and EPA, derived from fish. We therefore concluded it important to test whether the shorter chain ω-3 vegetable oil ALA also had antiarrhythmic effects, since this might also explain the beneficial effects seen on cardiovascular mortality in the Lyon Heart Study.

DETAILED DESCRIPTION:
Objective: We determined the effect of an ALA rich diet in reducing recurrence of atrial fibrillation as a further example of a cardiac arrhythmia.

Design: Randomized parallel design efficacy study. Setting: Three university hospital centers in the Bordeaux region, France. Patients: 98 successive patients successfully underwent electro cardioversion of whom 75 completed the study without major deviations according to the protocol.

Intervention: A canola margarine and oil together with a Mediterranean diet (ALA ω-3, 1.4 g/d) versus a conventional diet (control), with a one year follow-up.

Main outcome measure: Length of time to first recurrence of atrial fibrillation.

Significance: If ALA is antiarrhythmic this action may explain its cardioprotective effect in clinical trials and cohort studies.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in one of the three centers in the Bordeaux region, and who subsequently underwent successful electrocardioversion for atrial fibrillation.

Exclusion Criteria:

* included patients who were unable to receive electrocardioversion or those who were already enrolled in another trial
* patients who were unable or unwilling to comply with the diet recommendations (experimental or control) or follow-up requirements
* patients with clinically significant cardiac disease, advanced heart failure, cardiac cachexia, thyroid disease, treated or untreated, clinically significant hepatic or renal disease or a history of malignant disease or alcohol abuse were not included
* Taking ALA rich foods or recording intakes of ALA >2g/d on the control diet or reporting using <1g/d on the ALA diet was considered a major deviation from the protocol.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 1999-06; Study Completion 2003-06

PRIMARY OUTCOMES:
rate of recurrence and length of time to first recurrence of atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Renaud, MD, PhD, Principal Investigator — Emile Roux Hospital, A.P.H. Paris, 94456 Limeil-Brevannes, France
Locations (1):
- Emile Roux Hospital, Paris, France

REFERENCES:
- [Background] de Lorgeril M, Renaud S, Mamelle N, Salen P, Martin JL, Monjaud I, Guidollet J, Touboul P, Delaye J. Mediterranean alpha-linolenic acid-rich diet in secondary prevention of coronary heart disease. Lancet. 1994 Jun 11;343(8911):1454-9. doi: 10.1016/s0140-6736(94)92580-1. PMID 7911176